CLINICAL TRIAL: NCT04133350
Title: Patients With Heart Failure With Preserved Ejection Fraction Adherence to ASV Therapy Pilot Registry (PEP ASV Pilot Registry)
Brief Title: Patients With Heart Failure With Preserved Ejection Fraction Adherence to ASV Therapy (PEP ASV)
Acronym: PEP-ASV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to Recruit
Sponsor: Thomas Jefferson University (Other)
Collaborators: Inova Fairfax Hospital (Other); Heart and Diabetes Center North Rhine-Westphalia (Other); CLEMENS HOSPITAL (Unknown); Resmed Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19P.115
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Sleep Disorder; Breathing-Related; Heart Failure
MeSH Terms: conditions — Sleep Wake Disorders; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Patient Engagement (Experimental): All patients are enrolled into the Active Patient Engagement (APE) arm. This arm will receive the APE intervention.
  Interventions: Behavioral: Active Patient Engagement

INTERVENTIONS:
Behavioral: Active Patient Engagement — The APE intervention will be delivered through a patient-facing application and website called myAir, which provides patients with access to their own usage data, educational tips, and coaching.

SUMMARY:
This is a prospective, single-arm, unblinded pilot study and registry that aims to demonstrate adherence to adaptive servo-ventilation (ASV) therapy in patients with moderate to severe sleep disordered breathing who have been recently hospitalized. ASV therapy has been linked to improved outcomes in this population, but adherence to therapy is low. The AirCurve 10 ASV device that will be used for this study employs newer technologies, such as web-based monitoring and provides patients feedback, which may increase therapy adherence and therefore improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients 18 years or older 2. Patients with heart failure with preserved ejection fraction (HFpEF; LVEF ≥50%) 3. Hospital admission or equivalent (such as ER visit alone or clinic visit alone) and acute decompensated HF as determined by:

  1. Dyspnea at rest or with minimal exertion AND
  2. Treatment with at least one dose of IV diuretic or ultrafiltration AND
  3. At least two of the following signs and symptoms:

  i. Orthopnea ii. Pulmonary rales that do not clear with cough iii. Congestion on chest X-ray iv. Local BNP or NT pro-BNP level:
* No current AFib: BNP≥100 pg/mL or NT pro-BNP≥300 pg/mL OR
* Current AFib: BNP≥150 pg/mL or NT pro-BNP≥450 pg/mL 4. Sleep disordered breathing (SDB) documented by screening polygraphy with an AHI≥15 events/hour (e/hr) 5. Patient is able to fully understand study information and sign informed consent

Exclusion Criteria:

1. Right-sided heart failure without left-sided failure
2. Current chronic use (within 4 weeks of registry entry) of any PAP therapy (e.g., CPAP, APAP, or bi-level) or contraindicated for PAP therapy
3. Sustained systolic blood pressure <80 mmHg at baseline
4. Complex congenital heart disease
5. Constrictive pericarditis
6. Chronic hypoxemia as evidenced by sustained oxygen saturation ≤ 85% at rest during the day or at start of nocturnal oximetry recording or regular use of oxygen therapy (day or night)
7. Transient ischemic attack (TIA) or Stroke within 3 months prior to registry entry
8. Definite clinically evident acute myocardial infarction within 3 months of registry entry
9. Known amyloidosis, hypertrophic obstructive cardiomyopathy, or arteriovenous fistulas
10. Moderate or greater valvular heart disease as the primary reason for heart failure
11. In the opinion of the investigator, the index acute decompensated HF event was not due primarily to uncontrolled AFib with fast ventricular response rate
12. Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Adherence (hours/night) | 3 months
  Demonstrate acceptable adherence to ASV therapy can be achieved in patients with moderate to severe SDB in a recently hospitalized population of Heart Failure patients with preserved ejection fraction (HFpEF).

SECONDARY OUTCOMES:
Quality of Life Score - | 3 months
  Quality of life will be assessed using the KCCQ-12, a 12-item validated instrument that measures Quality of Life in heart failure patients on a scale of 0-100. Higher scores indicate higher Quality of Life

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - INOVA (Inova Heart and Vascular Institute, Inova Fairfax Hospital), Falls Church, Virginia
- Germany (2):
  - Herz- und Diabeteszentrum, Nordrhein-Westfalen, Bad Oeynhausen, Ruhr-Universität Bochum
  - Ludgerus Clinic, Department of Cardiology, Clemens Hospital, Münster

IPD SHARING:
Plan to Share IPD: Undecided